CLINICAL TRIAL: NCT03447600
Title: The Impact of Weight Loss Through Alternate Day Fasting on Homeostatic and Hedonic Appetite Control and Eating Behaviour: a Proof of Concept Randomized Controlled Trial
Brief Title: Diet-Induced Variability in Appetite (DIVA)
Acronym: DIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Dr Graham Finlayson, Chair in Psychobiology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LDS-DIVA-2017
Record Dates: First submitted 2018-02-09; First posted 2018-02-27 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternate day fasting (Experimental): Participants randomised to Alternate Day Fasting weight loss intervention. One day fasting of 25% total energy requirements alternated with one day ad libitum intake until study completion at >/=5% weight loss which is an average of 12 weeks.
  Interventions: Behavioral: Alternate Day Fasting
- Continuous caloric restriction (Active Comparator): Participants randomised to continuous caloric restriction weight loss intervention. Every day intake of 75% total energy requirements until study completion at >/=5% weight loss which is an average of 12 weeks.
  Interventions: Behavioral: Continuous dietary restriction

INTERVENTIONS:
Behavioral: Alternate Day Fasting — 25% daily energy requirements every other day until study completion at >/=5% weight loss which is an average of 12 weeks.
  Arms: Alternate day fasting
Behavioral: Continuous dietary restriction — 25% daily energy requirements every other day until study completion at >/=5% weight loss which is an average of 12 weeks.
  Arms: Continuous caloric restriction

SUMMARY:
The aim of this study is to test the hypothesis that dietary weight loss (WL) through alternate day fasting (ADF) will enhance appetite control, health markers and wellbeing following WL compared to standard daily calorie restriction (CR).

DETAILED DESCRIPTION:
This is a proof of concept randomized controlled trial in which overweight/obese females will be randomised to a dietary weight loss intervention (ADF or CR) to achieve ≥5% WL. Behavioural measures of appetite control including ad libitum intake after a fixed meal, body composition, resting metabolic rate, measured physical activity and daily energy expenditure, sleep quality, hedonic food reward and eating behaviour traits will be assessed before, during and after the WL intervention in those who reach the target weight loss within 12 weeks. After weight loss phase, participants will be given standard healthy eating and physical activity advice for weight maintenance and body weight will be followed up after weight loss at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged between 18 and 55 years at the time of signing informed consent
* BMI of 25.0 - 34.9 kg/m2

Exclusion Criteria:

* Significant health problems which in the opinion of the investigator, might jeopardise participant's safety or compliance with the protocol
* Currently enrolled in a weight loss programme or following a specific diet plan.
* History of eating disorders including binge eating.
* Taking any medication or supplements known to affect appetite or weight within the past month and/or during the study
* Pregnant, planning to become pregnant or breastfeeding
* History of anaphylaxis to food
* Known food allergies or food intolerance
* Smokers and those who have recently ceased smoking (< 6 months)
* BMI < 24.9 kg/m2 or > 35 kg/m2
* Volunteers having lost significant amount of weight in the previous 6 months (± 4kg)
* Volunteers who exercise > 3 days per week or have significantly changed their physical activity patterns in the past 6 months or who intend to change them during the study
* Participants receiving systemic or local treatment likely to interfere with evaluation of the study parameters
* Participants who work in appetite or feeding related areas.
* Participants who do shift work

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Change in energy intake from ad libitum lunch | week 0, week 3 and at study completion, an average of 12 weeks
  Measured changes in ad-libitum energy intake following consumption of formulated test meal in comparison to control

SECONDARY OUTCOMES:
Change in Visual Analogue Scale (VAS) ratings of appetite | week 0, week 3 and at study completion, an average of 12 weeks
  Change in ratings of hunger, satiety, fullness and prospective food consumption before, after and between meals. Scale range is minimum 0 to maximum 100mm. A composite appetite score will be calculated from the average of scores on hunger, satiety, fullness and prospective food consumption scales. A higher score is considered a worse outcome.
Change in Control of Eating Questionnaire (CoEQ) scale scores | week 0, week 3 and at study completion, an average of 12 weeks
  21-item scale; subscales are average of relevant items; subscales are computed for dimensions of Craving Control, Craving for Savoury, Craving for Sweet, Positive Mood; minimum subscale score = 0, maximum subscale score = 100; higher values are better outcome for Craving Control and Positive Mood subscales; lower values are better outcome for Craving for Sweet and Craving for Savoury subscales.
Change in explicit liking of food from Leeds Food Preference Questionnaire | week 0, week 3 and at study completion, an average of 12 weeks
  Leeds Food Preference Questionnaire is a computer-based task with subscales scores for the 4 food categories high fat and sweet, high fat and non-sweet, low fat and sweet and low fat and non-sweet (minimum score = 0, maximum score = 100), Higher values for high fat food categories relative to low fat food categories considered worse outcome.
Change in explicit wanting of food from Leeds Food Preference Questionnaire scores | week 0, week 3 and at study completion, an average of 12 weeks
  Leeds Food Preference Questionnaire is a computer-based task with subscales scores for the 4 food categories high fat and sweet, high fat and non-sweet, low fat and sweet and low fat and non-sweet (minimum score = 0, maximum score = 100), Higher values for high fat food categories relative to low fat food categories considered worse outcome.
Change in relative preference of food from Leeds Food Preference Questionnaire scores | week 0, week 3 and at study completion, an average of 12 weeks
  Leeds Food Preference Questionnaire is a computer-based task with subscales scores for the 4 food categories high fat and sweet, high fat and non-sweet, low fat and sweet and low fat and non-sweet (minimum score = 0, maximum score = 48), Higher values for high fat food categories relative to low fat food categories considered worse outcome.
Change in implicit wanting of food from Leeds Food Preference Questionnaire scores | week 0, week 3 and at study completion, an average of 12 weeks
  Leeds Food Preference Questionnaire is a computer-based task with subscales scores for the 4 food categories high fat and sweet, high fat and non-sweet, low fat and sweet and low fat and non-sweet (minimum score = -100, maximum score = 100), Higher values for high fat food categories relative to low fat food categories considered worse outcome.
Change in VAS rating of palatability post lunch | week 0, week 3 and at study completion, an average of 12 weeks
  Change in ratings of pleasantness, desire to eat more and palatability after the lunch test meal
Change in fat mass | week 0, week 3 and at study completion, an average of 12 weeks
  Change in fat mass from iDXA/BodPod
Change in fat free mass | week 0, week 3 and at study completion, an average of 12 weeks
  Change in fat free mass from iDXA/BodPod
Change in resting metabolic rate | week 0, week 3 and at study completion, an average of 12 weeks
  Change in resting metabolic rate from indirect calorimetry
Change in free-living physical activity | week 0, week 3 and at study completion, an average of 12 weeks
  Change in 7-day free-living physical activity from SenseWear Armband

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Beaulieu, PhD, Principal Investigator — University of Leeds; Graham Finlayson, PhD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beaulieu K, Casanova N, Oustric P, Turicchi J, Gibbons C, Hopkins M, Varady K, Blundell J, Finlayson G. Matched Weight Loss Through Intermittent or Continuous Energy Restriction Does Not Lead To Compensatory Increases in Appetite and Eating Behavior in a Randomized Controlled Trial in Women with Overweight and Obesity. J Nutr. 2020 Mar 1;150(3):623-633. doi: 10.1093/jn/nxz296. PMID 31825067